CLINICAL TRIAL: NCT05997953
Title: Assessment of the Edinburgh Postnatal Depression Scale as Screening Tool for Postpartum Depression Among Women Delivering at Egyptian Tertiary Care System University Hospital: Prevalence and Risk Factors Analysis
Brief Title: Screening of Postpartum Depression in Egyptian Women
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Other Study IDs: 520235
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Edinburgh Postnatal Depression Scale — Edinburgh Postnatal Depression Scale used as screening tool for postpartum depression

SUMMARY:
The goal of this cross-sectional study is to assess the Edinburgh Postnatal Depression Scale as screening tool for Postpartum Depression among women delivering at Egyptian tertiary health care system, University Hospital, regarding Prevalence and risk factors.

participants of this study with fill the Edinburgh Postnatal Depression Scale and their socio-demographic, obstetric and psychological data will be collected and analysed.

prevalence of postpartum depression in Egyptian women will be assessed as well as the associated risk factors

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent vaginal/cesarean delivery and reported for follow and willing to participate in the study.

Exclusion Criteria:

* Patients who were unwilling to participate in the study.
* Patients who are having difficulties comprehending the questionnaire of the study.
* Women who were on psychiatric medication during pregnancy.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: 2000 patients who underwent either vaginal birth or cesarean section at El-Hussien University Hospital and agreed for followup and participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Number screening positive for possible postpartum depression by Arabic EPDS | 2 weeks postpartum
  Number of participants screening positive for possible postpartum depression, defined as a score of 13 or higher on the validated Arabic version of the Edinburgh Postnatal Depression Scale (EPDS) Participants with a positive screen (EPDS score ≥13) will be referred for psychiatric consultation for diagnostic confirmation and treatment of postpartum depression

SECONDARY OUTCOMES:
Sociodemographic, clinical, and psychosocial predictors of postpartum depression risk | At 2 weeks postpartum
  Identification of sociodemographic, clinical, and psychosocial risk factors associated with screening positive for possible postpartum depression, as determined by bivariate and multivariate regression analyses of factors correlated with an Arabic EPDS score ≥13.
  Sociodemographic factors will include maternal age, education level, occupation, socioeconomic status, etc.
  Clinical factors will include obstetric history, delivery method, neonatal health status, etc.
  Psychosocial factors will include social support, stress levels, family dynamics, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty od Medicine, Department of Obstetrics and Gynecology., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No